CLINICAL TRIAL: NCT02791737
Title: Maintaining Fitness: Exercise in Patients With Hematologic Malignancy
Brief Title: Exercise Prehab in Older Adults With Hematologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Ashley Rosko, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-16016; NCI-2016-00446 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
Keywords: Hematologic Malignancy; Exercise; Decreased Physical Activity
MeSH Terms: conditions — Hematologic Neoplasms; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (otago exercise programme) (Experimental): Patients attend 8 physical therapy visits twice monthly for 4 months or until transplant. Patients also undergo an individualized exercise program at home for 6 months. The program comprises 3 main components: walking over 30 minutes twice a week, strengthening and balance retraining exercise over 30 minutes three times a week.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Procedure: Physical Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Complete individualized exercise program
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Physical Therapy — Complete individualized exercise program
  Other Names: Physiatric Procedure; Physical Medicine Procedure; Physical Therapeutics; Physical Therapy Procedure; Physiotherapy; Physiotherapy Procedure; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot trial studies a structured exercise program intervention in improving physical activity in older patients with hematologic malignancies undergoing cancer therapy. Patients with hematologic malignancies are at an increased risk of functional dependence and injury. Structured exercise programs, such as the Otago exercise programme (OEP), may improve balance, strength, and prevent fall-related injury in older patients with hematologic malignancies undergoing cancer therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of implementing a structured exercise program by evaluating recruitment and retention, exercise program adherence, sustainability, adverse events, and implementation challenge.

SECONDARY OBJECTIVES:

I. To calculate preliminary effect sizes of the impact of an exercise program in patients with hematologic malignancy undergoing therapy, as measured by:

* Cancer and Aging Research Group (CARG) Geriatric Assessment Tool parameters.
* Change in Short Physical Performance Battery (SPPB).
* Number and severity of falls.
* Impact of motivation and self-efficacy on adherence.
* Hospital readmission rates (if applicable).
* Length of inpatient stays (if applicable).
* Patient Reported Outcome Measurement Information System (PROMIS) for Health related quality of life (HRQL).
* Correlative analysis of peripheral blood biomarkers of aging and inflammation (cyclin-dependent kinase inhibitor 2A [p16], inflammatory biomarkers, immunosenescence, micro [mi] ribonucleic acid [RNA]).

OUTLINE:

Patients attend 8 physical therapy visits twice monthly for 4 months or until transplant. Patients also undergo an individualized exercise program at home for 6 months. The program comprises 3 main components: walking over 30 minutes twice a week, strengthening and balance retraining exercise over 30 minutes three times a week.

After completion of study, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancy receiving care (chemotherapy, immunotherapy, targeted agents, bone marrow transplant, or other) for their hematologic malignancy at the Ohio State University
* Impairments in physical function, as defined by a score < 9 on the SPPB pre-screen
* Medical clearance from an oncologist or primary care physician stating the participant is able to participate in an unsupervised, moderate-intensity physical activity program
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prisoners
* Any medical condition including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study procedures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Rosko, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Rosko A, Huang Y, Jones D, Presley CJ, Jaggers J, Owens R, Naughton M, Krok-Schoen JL. Feasibility of implementing an exercise intervention in older adults with hematologic malignancy. J Geriatr Oncol. 2022 Mar;13(2):234-240. doi: 10.1016/j.jgo.2021.07.010. Epub 2021 Aug 24. PMID 34446377
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited from the hematology clinics at The Ohio State University Comprehensive Cancer Center August 2016 to January 2018.
Period: Overall Study
Arm/Group | Supportive Care (Otago Exercise Programme)
Started | 30 (Consented to enrollment)
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 30
Age, Customized [Median (Full Range); unit: years] | 75.5 [62 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AE), Graded According to Common Terminology Criteria for Adverse Events Version 5.0
Description: Adverse Events and their severity will be captured and graded according to Common Terminology Criteria for Adverse Events Version 5.0, and whether any events can be attributed to exercise.
Time Frame: Study Visit 1 (Baseline) Study Visit 2 (4 months) Study Visit 3 (6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 30
Participants | 0

2. Primary Outcome: Percentage of Eligible Patients Completing the OEP
Description: Feasibility defined as 80% of eligible of patients completing the OEP. The proportion of screened patients who agree to participate, the proportion of patients who attend certain percentage of assigned physical therapy (PT) sessions and the proportion of patients who complete the whole study along will be described with respective 95% confidence intervals. Study implementation and challenges will be evaluated by patient exercise logs. Exercise levels at home will also be assessed by exercise diary log
Time Frame: Study Visit 1 (Baseline) Study Visit 2 (4 months) Study Visit 3 (6 months)
Measure: Number; unit: percent of patients
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 30
percent of patients | 66.7

3. Secondary Outcome: Biomarker Expression Levels
Description: Specific biomarkers of aging will be explored to determine a relationship with molecular markers of aging and epigenetic age with a frailty phenotype. mRNA isolates will be analyzed using a nanostring codeset. The regulation levels of killer cell immunoglobulin-like receptors (KIRs) will be reported. Both KIR_Activating_Subgroup_1 and KIR_Activating_Subgroup_2 levels will be reported. Participants are classified based on a frailty scale: favorable (fit patients based on frailty scale), mid (intermediately fit), unfavorable (frail). Negative values indicate a downregulation of gene expression and positive values indicate an upregulation of gene expression.
Time Frame: Study Visit 1 (Baseline), and study visit 3 (6 months)
Population: number analyzed is the number of patients that fit into each category: unfavorable, mid, and favorable.
Measure: Median (Full Range); unit: cycle threshold
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 26
cycle threshold
  KIR_Activating _Subgroup_1 Unfavorable median: number analyzed (Participants) | 10
  KIR_Activating _Subgroup_1 Unfavorable median | 1.26 [-0.42 to 2.33]
  KIR_Activating _Subgroup_1 Mid median | -0.19 [-2.69 to 2.79]
  KIR_Activating _Subgroup_1 Favorable median: number analyzed (Participants) | 10
  KIR_Activating _Subgroup_1 Favorable median | 0.15 [-0.42 to 2.33]
  KIR_Activating_Subgroup_2 Unfavorable median: number analyzed (Participants) | 10
  KIR_Activating_Subgroup_2 Unfavorable median | 0.62 [-0.54 to 1.20]
  KIR_Activating _Subgroup_2 Mid median | -0.05 [-2.82 to 1.18]
  KIR_Activating _Subgroup_2 Favorable median: number analyzed (Participants) | 10
  KIR_Activating _Subgroup_2 Favorable median | 0.20 [-0.54 to 1.86]

4. Secondary Outcome: Change in Geriatric Assessment (GA) Measured Using The Cancer and Aging Research Group (CARG) Geriatric Assessment (G)A-patient Reported Karnofsky Performance Status (KPS) for Patients Undergoing Transplant
Description: Patient-reported KPS31 measures the patients self-reported level of physical function. Scoring extends from 30 (severely disabled) - 100 (normal), with a higher score indicating a higher level of physical function. Descriptive statistics of these measurements will be provided as well as graphs in order to help visualize the change over time.
Time Frame: Study Visit 1 (Baseline) Study Visit 2 (4 months) Study Visit 3 (6 months)
Population: only 7 patients had transplants
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 7
score on a scale
  Visit 1 | 80 [40 to 100]
  Visit 2: number analyzed (Participants) | 6
  Visit 2 | 85 [60 to 100]
  Visit 3: number analyzed (Participants) | 5
  Visit 3 | 90 [60 to 100]

5. Secondary Outcome: Change in Geriatric Assessment (GA) Measured Using the CARG GA-patient Reported Karnofsky Performance Status (KPS)
Description: as for outcome 4
Time Frame: Study Visit 1 (Baseline) Study Visit 2 (4 months) Study Visit 3 (6 months)
Population: Patients did not complete all visits
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 30
score on a scale
  Visit 1 | 80 [40 to 100]
  Visit 2: number analyzed (Participants) | 23
  Visit 2 | 90 [60 to 100]
  Visit 3: number analyzed (Participants) | 20
  Visit 3 | 90 [50 to 100]

6. Secondary Outcome: Health Related Quality of Life (HRQL) Measured Using the PROMIS
Description: Patient-Reported Outcome Measurement Information System (PROMIS) Global Health Scale Short Form v1.1 HRQL measures provide information to the clinician regarding the patient experience of treatment or intervention. The PROMIS Global Health Scale has been rigorously tested for reliability and validity and can be applied to all populations, where higher scores reflect improved quality of life. It consists of 10 questions and was given to the patients for self-administration at three intervals. Descriptive statistics of these measurements will be provided as well as graphs in order to help visualize the change over time. 5 point Likert scale higher values represent a better quality of life. PROMIS scores, developed by the NIH, are usually presented as T-scores, where the average score is 50 and a standard deviation is 10.
Time Frame: Study visit 1 (Baseline), Study visit 2 (month 4), and study visit 3 (month 6, completion of study)
Population: Patients did not complete all visits
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 30
score on a scale
  Visit 1 | 32.4 [19.9 to 47.7]
  Visit 2: number analyzed (Participants) | 23
  Visit 2 | 34.9 [26.7 to 47.7]
  Visit 3: number analyzed (Participants) | 20
  Visit 3 | 36.2 [19.9 to 47.7]

7. Secondary Outcome: Change in HRQL Measured Using the PROMIS for Patients Undergoing Transplant
Description: as for outcome 6
Time Frame: Study Visit 1 (Baseline) Study Visit 2 (4 months) Study Visit 3 (6 months)
Population: only 7 patients received transplants
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 7
score on a scale
  Visit 1 | 34.9 [23.5 to 47.7]
  Visit 2: number analyzed (Participants) | 6
  Visit 2 | 36.2 [29.6 to 42.3]
  Visit 3: number analyzed (Participants) | 5
  Visit 3 | 34.9 [32.4 to 39.8]

8. Secondary Outcome: Number of Falls (Inpatient and Outpatient)
Description: The total number of falls experienced by participants will be reported. Both falls that occur inpatient and outpatient will be included.
Time Frame: Up to 6 months
Measure: Number; unit: number of falls
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 30
number of falls | 3

9. Secondary Outcome: Change in Physical Performance Measured Using the Short Physical Performance Battery (SPPB)
Description: Scores are assigned for each of the tests and an aggregate score is assigned ranging from 0-12, with higher scores indicating greater physical function. SPPB scores are classified into 4 categories: very low physical function (0-3); low physical function (4-6); moderate physical function (7-9) and high physical function (10-12). An alpha internal consistency of 0.76 has been reported
Time Frame: Study Visit 1 (Baseline) Study Visit 2 (4 months) Study Visit 3 (6 months)
Population: Patients did not complete all visits
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 30
units on a scale
  Visit 1 | 7 [0 to 11]
  Visit 2: number analyzed (Participants) | 23
  Visit 2 | 11 [4 to 12]
  Visit 3: number analyzed (Participants) | 20
  Visit 3 | 9 [2 to 12]

10. Secondary Outcome: Change in Physical Performance Measured Using the SPPB for Patients Undergoing Transplant
Description: as for outcome 9
Time Frame: Study Visit 1 (Baseline) Study Visit 2 (4 months) Study Visit 3 (6 months)
Population: only 7 patients received transplant
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 7
units on a scale
  Visit 1 | 8 [0 to 10]
  Visit 2: number analyzed (Participants) | 6
  Visit 2 | 11.5 [10 to 12]
  Visit 3: number analyzed (Participants) | 5
  Visit 3 | 10 [2 to 12]

11. Secondary Outcome: Percentage of Patients With Hospital Readmission for Patients Undergoing Transplant
Description: Evaluating the frequency (percentage of patients with hospital re-admissions) within 90 days
Time Frame: At 90 days
Measure: Number; unit: percentage of patients
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 7
percentage of patients | 42.9

12. Secondary Outcome: Length of Inpatient Stays for Patients Undergoing Transplant
Description: Descriptive statistics of these measurements will be provided as well as graphs in order to help visualize the change over time. The proportion of patients who achieve meaningful change in these scores will be described with 95% confidence intervals. Difference from baseline will be tested with Wilcoxon signed rank test or McNemar's test for continuous or categorical variables respectively.
Time Frame: Up to 6 months
Measure: Median (Full Range); unit: days
Arm/Group | Supportive Care (Otago Exercise Programme)
Number analyzed (Participants) | 3
days | 18 [16 to 18]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected for patients from baseline through study completion utilizing the CTCAE version 5.0 to determine the severity of the reaction for adverse event reporting from baseline to after study completion an average of 1 year.
Arm/Group | Supportive Care (Otago Exercise Programme)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT02791737/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT02791737/ICF_001.pdf